CLINICAL TRIAL: NCT00800007
Title: A Phase 1/2 Randomized, Placebo-Controlled, Double-Blind, Dose-Escalation Study to Evaluate the Safety, Tolerability, and Pharmacodynamics of Multiple Intravenous Doses of ANZ-521 in Hepatitis C Patients
Brief Title: Study of Safety and Tolerability of Multiple Intravenous Doses of ANZ-521 in Adults With Chronic Hepatitis C Virus
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Anza Therapeutics, Inc. (Industry)
Responsible Party: Dung Thai, MD, PhD/Chief Medical Officer, Anza Therapeutics, Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ANZ-521-101
Record Dates: First submitted 2008-11-26; First posted 2008-12-01 (Estimated); Last update posted 2009-02-20 (Estimated); Status verified 2009-02

CONDITIONS: Chronic Hepatitis C
Keywords: Hepatitis C, HCV, ANZ-521, Listeria
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ANZ-521 (Active Comparator)
  Interventions: Drug: ANZ-521
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ANZ-521 — 3x10^7 cfu or 3x10^8 cfu ANZ-521 in 250 mL, IV over 2 hours, every 28 days for up to 3 doses.
  Arms: ANZ-521
Drug: Placebo — 250 mL normal saline, IV over 2 hours, every 28 days for up to 3 doses.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, immunogenicity, and antiviral effects of multiple intravenous doses of ANZ-521 in patients with chronic Hepatitis C virus.

DETAILED DESCRIPTION:
This Phase 1/2 Randomized, Placebo Controlled, Double-Blind clinical trial will evaluate the safety, tolerability, and pharmacodynamics of ANZ-521, an investigational product that is a weakened form (attenuated) of Listeria monocytogenes, a type of bacteria that is commonly found in the environment. ANZ-521 has been altered in the lab to reduce its ability to cause disease, while maintaining stimulation of the immune system. ANZ-521 has also been genetically modified with recombinant DNA to encode consensus sequence antigens called NS5B polymerase and NS3 proteinase that correspond to viral proteins found on the virus causing Hepatitis C. It is hoped that ANZ-521 will stimulate an immune response to the Hepatitis C virus (HCV) in the liver, thereby demonstrating an effective therapy for individuals with chronic HCV infection.

The purpose of this first clinical trial with ANZ-521 is to identify an appropriate dose of the investigational agent for later clinical studies and to explore safety when given to consenting adults with HCV. Immunological response to ANZ-521 in study participants will also be measured. Patients who choose to enter the study must meet all study entry criteria. The first part of the study (Part A) will enroll subjects who have received prior treatment with standard of care therapy for HCV. The second part of the study (Part B) will enroll subjects who have not previously received standard of care therapy for HCV or were intolerant to standard of care. Qualifying study patients will be assigned to receive one of at least 2 dose levels of ANZ-521 or placebo. Each patient may receive up to 3 intravenous administrations (28 days apart) of ANZ-521 or placebo at their assigned dose level.

ELIGIBILITY:
Inclusion Criteria:

* Chronic liver disease consistent with chronic hepatitis C infection, genotype 1, for at least 6 months
* For Part A only: patients who have had a full course of interferon and ribavirin as defined by the NIH Consensus Statement for the Management of Hepatitis C: 2002 (Management of hepatitis C: 2002, 2002) and have a detectable viral titer at Screening.
* For Part B only: patients who are HCV treatment-naïve with known contraindications (i.e., history of depression) to interferon and ribavirin combination therapy; patients who have started on interferon and ribavirin but stopped therapy early due to intolerance; patients who have not received interferon and ribavirin and have refused therapy
* Plasma HCV RNA viral titer of ≥ 2 logs above the assay cutoff measured at Screening.
* Females must be of non-child bearing potential [i.e., 1 year post menopausal or documented as being surgically sterile].
* Men must agree to use an acceptable form of birth control through the study and for 28 days after final dose of ANZ-521.
* Liver biopsy within the last 3 years with an Ishak Score <3 of FibroSURE test score <0.59.
* Compensated liver disease (Child-Pugh class A) with the adequate organ function as defined by study-specific laboratory tests.
* Signed Informed Consent and willing and able to comply with all study procedures.

Exclusion Criteria:

* Patients who are null responders to interferon-based therapy as defined by a less than 1-log decrease in viral titer from baseline during treatment.
* Treatment with anti-HCV therapy within one month prior to study.
* History of infection with Listeria.
* History of having received an experimental HCV vaccine (therapeutic or preventive).
* Known allergy to both penicillin and sulfa drugs, or component of the study drug product (e.g., glycerol).
* Current or prior history of certain study-specified heart, liver, kidney, lung, neurological, immune or other medical condition.
* Artificial (prosthetic) joint or other artificial implant or devices that cannot be easily removed.
* History of malignancy of any type, other than surgically excised non-melanomatous skin cancers or in situ cervical cancer within 5 years.
* Taking certain medications such as more than 2 g of acetaminophen per day, systemic antibiotics within 14 days of study entry, another investigational product within 28 days of study entry.
* Recent hospitalization or planned surgery requiring general anesthesia or sedation.
* Drug screen positive for cocaine.
* Positive for HIV or Hepatitis B antibodies.
* Blood donation of more than 450 mL within 8 weeks of study entry.
* Other condition that might affect the subject's ability to give informed consent or comply with study requirements.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2008-11; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Subject incidence of AEs, clinically relevant changes in lab values, ECGs, and vital signs | 84 days

SECONDARY OUTCOMES:
Plasma HCV RNA titers relative to baseline | 84 days
Serum transaminase levels relative to baseline | 84 days
Innate and adaptive immune responses induced by ANZ-521 | 84 days
Blood, stool, and urine cultures of ANZ-521 | 84 days

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Advanced Clinical Research Institute, Anaheim, California
  - Alamo Medical Research, San Antonio, Texas